CLINICAL TRIAL: NCT03928509
Title: Cohort as Part of Undergraduate Medical Studies at the University of Sherbrooke
Status: Recruiting | Type: Observational
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Sponsor
Other Study IDs: MP-31-2019-3172
Record Dates: First submitted 2019-03-06; First posted 2019-04-26 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Public Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Estrie CIUSSS: Subjects from the Estrie's Integrated Health and Social Services Centre
  Interventions: Other: No intervention
- Saguenay-Lac-Saint-Jean CIUSSS: Subjects from the Saguenay-Lac-Saint-Jean's Integrated Health and Social Services Centres
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The main goals of this project are to support the research training of undergraduate medical students at the University de Sherbrooke and promote planning of health services a better knowledge of the prevalence, social, and geographic distribution of public health issues in several regions in Quebec.

To meet the objectives of the project, a population-based prospective study linked to several regions in Quebec public health surveys is proposed.

Monitoring and data collection will be provided by 3rd year undergraduate medical students at University de Sherbrooke through telephone interviews.

The research themes will be proposed by various researchers affiliated with the University de Sherbrooke. They will be selected yearly by an internal scientific committee and included in the questionnaires administered by the students.

ELIGIBILITY:
Inclusion criteria:

* Participants will have been diagnosed with covid-19 between November 2020 and May 2021;
* Place of residence: province of Quebec.

Exclusion criteria :

- Unfit adults.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population is everyone who has been diagnosed with covid-19 in several regions in Quebec
Sampling Method: Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2019-08-29 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Health questionnaire | Once a year through study completion.
  General health questionnaire including questions about lifestyle, access to health services, comorbidities, mental health, alcohol and drugs consumption. Additional questions regarding more specific themes (Lyme disease, medical aid in dying, COVID-19, etc.) will be added or adapted yearly.
  Most of the questions are individually based on previously accepted or previously used questionnaires and thus, the health questionnaire used in this project does not include a specific scale of measurement for each subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Farand, MD MSc, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre Hospitalier Universitaire de Sherbrooke, departement de médecine, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes